CLINICAL TRIAL: NCT04628377
Title: Prognostic Implication of Angiography-Derived Index of Microcirculatory Resistance in Successfully Reperfused STEMI Patients
Brief Title: Prognostic Implication of Angiography-Derived IMR in STEMI Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: RainMed Medical Group (Industry)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant Professore, Samsung Medical Center
Other Study IDs: NCTSTEMI2575
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Acute ST-segment Elevation Myocardial Infarction
Keywords: STEMI; Index of microcirculatory resistance; Quantitative flow ratio; Fractional flow reserve; Prognosis; Angiography-derived IMR
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnostic Accuracy Cohort: Patients are subgroup of previously published study (JACC Cardiovascular Intervention 2020;13:1155-67), which evaluated invasive physiologic indices from culprit and non-culprit vessels of acute myocardial infarction patients. From the study cohort, 31 STEMI patients who underwent IMR measurement in culprit vessel after successful revascularization will be analyzed. In these patients, diagnostic accuracy of angiography-derived IMR will be compared with invasive IMR.
  Interventions: Device: Angiography-drived Index of Microcirculatory Resistance
- Prognosis Cohort: Prognosis cohort, in which angiography-derived IMR will be measured in the culprit vessel after successful revascularization. Those patients have follow-up data after 10 years from index procedure. This cohort is STEMI subgroup derived from Institutional registry of Samsung Medical Center, whose results were previously published (JACC Cardiovascular Intervention. 2019 Apr 8;12(7):607-620.) Among 490 STEMI patients from the overall study cohorts, 309 patients with available angiograms and who were suitable for angiographic FFR and IMR measurement will be analyzed. Primary clinical outcome will be cardiac death at 10 years from index procedure. Secondary outcome will be any myocardial infarction, ischemia-driven revascularization, definite or probable stent thrombosis, congestive heart failure admission at 10 years from index procedure.
  Interventions: Device: Angiography-drived Index of Microcirculatory Resistance

INTERVENTIONS:
Device: Angiography-drived Index of Microcirculatory Resistance — From coronary angiographic images, angiography-derived IMR will be calculated based on mathematical calculation.
  Angiography-derived IMR = (hyperemic Pa x angiography-derived FFR) x (vessel length / {K x V diastole}).
  Hyperemic Pa will be estimated from resting Pa according to prespecified equation.
  Other Names: Angiography-derived IMR

SUMMARY:
Coronary microcirculatory dysfunction has been known to be prevalent even after successful revascularization of STEMI patients. Previous study presented that index of microcirculatory resistance (IMR) in culprit vessel of STEMI patients showed significant association with the risk of cardiac death or heart failure admission. Recent technical development enabled angiographic derivation of IMR without pressure wire, hyperemic agents, or theromdilution method. In this regard, the current study will evaluate prognostic implication of angiography-derived IMR in STEMI patients who were successfully revascularized.

DETAILED DESCRIPTION:
Coronary microcirculatory dysfunction has been known to be prevalent even after successful revascularization of STEMI patients. Previous study presented that index of microcirculatory resistance (IMR) in culprit vessel of STEMI patients showed significant association with the risk of cardiac death or heart failure admission. Recent technical development enabled angiographic derivation of IMR without pressure wire, hyperemic agents, or theromdilution method. In this regard, the current study will evaluate prognostic implication of angiography-derived IMR in STEMI patients who were successfully revascularized.

The study cohorts consist with 2 separate cohort: first, diagnostic accuracy cohort, which will evaluate diagnostic accuracy of angiography-derived IMR for invasive IMR. For this, 31 patients with culprit vessel IMR measurement at the time of primary PCI will be evaluated. The patients cohort is the subgroup of previous registry (NCT02186093). Second, prognosis cohort, in which angiography-derived IMR will be measured in the culprit vessel after successful revascularization. Those patients have follow-up data after 10 years from index procedure. This cohort is STEMI subgroup derived from Institutional registry of Samsung Medical Center, whose results were previously published (JACC Cardiovascular Intervention. 2019 Apr 8;12(7):607-620.) Among 490 STEMI patients from the overall study cohorts, 309 patients with available angiograms and who were suitable for angiographic FFR and IMR measurement will be analyzed. Primary clinical outcome will be cardiac death at 10 years from index procedure. Secondary outcome will be any myocardial infarction, ischemia-driven revascularization, definite or probable stent thrombosis, congestive heart failure admission at 10 years from index procedure.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients who were successfully revascularized for culprit vessel
* analyzable angiograms at the index procedure

Exclusion Criteria:

* Previous coronary artery bypass grafting
* Coronary bypass graft as culprit vessel
* Patients with unclear culprit vessel
* limited image quality of coronary angiography
* Insufficient angiographic project for TIMI frame count
* Severe tortuosity of culprit vessel
* No optimal projection for reconstruction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnostic Accuracy Cohort 31 STEMI patients who underwent IMR measurement in culprit vessel.
  Prognosis Cohort 309 patients with available angiograms and who were suitable for angiographic FFR and IMR measurement and have 10 years follow-up data.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2003-05-26 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | at the index procedure
  Diagnostic accuracy of angiography-derived IMR to predict invasive IMR
Cardiac death or heart failure admission | at 10 years from index procedure
  Cardiac death or heart failure admission

SECONDARY OUTCOMES:
Any myocardial infarction | at 10 years from index procedure
  Any myocardial infarction
Ischemia-driven revascularization | at 10 years from index procedure
  Ischemia-driven revascularization
Stent thrombosis | at 10 years from index procedure
  Definite or probable stent thrombosis according to ARC definition
Congestive heart failure admission | at 10 years from index procedure
  Admission for congestive heart failure
Major adverse cardiac events | at 10 years from index procedure
  a composite of cardiac death, any myocardial infarction, ischemia-driven revascularization, definite or probable stent thrombosis, or congestive heart failure admission
Cardiac death | at 10 years from index procedure
  Cardiac death
All-cause death | at 10 years from index procedure
  All-cause death
Heart failure admission | at 10 years from index procedure
  Heart failure admission

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized study data can be shared upon reasonable proposition. Principle investigator will review the request and decide whether the study data will be shared.

REFERENCES:
- [Derived] Choi KH, Dai N, Li Y, Kim J, Shin D, Lee SH, Joh HS, Kim HK, Jeon KH, Ha SJ, Kim SM, Jang MJ, Park TK, Yang JH, Song YB, Hahn JY, Doh JH, Shin ES, Choi SH, Gwon HC, Lee JM. Functional Coronary Angiography-Derived Index of Microcirculatory Resistance in Patients With ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Interv. 2021 Aug 9;14(15):1670-1684. doi: 10.1016/j.jcin.2021.05.027. PMID 34353599